CLINICAL TRIAL: NCT01085188
Title: Effectiveness of Assertive Continuing Care for Youth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Mark D. Godley, Ph.D./Director of Research and Development, Chestnut Health Systems
Allocation: Randomized | Model: Factorial | Purpose: Treatment
Other Study IDs: 1018-1201
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

ARMS (4):
- Assertive Continuing Care (ACC) (Experimental): Behavioral intervention comprised of the community reinforcement approach plus case management delivered in home and other community settings to youth and their caregivers.
  Interventions: Behavioral: ACC; Behavioral: UCC
- Contingency Management (CM) (Experimental): Using a prize drawing system (no, low, medium and large value prizes) with adolescents could earn escalating prize drawing opportunities by completing verifiable pro-social activities and providing negative urine test and breath alcohol test results.
  Interventions: Behavioral: CM; Behavioral: UCC
- ACC + CM (Experimental): This arm is the combination of arms 1 and 2.
  Interventions: Behavioral: ACC; Behavioral: CM; Behavioral: UCC
- Usual Continuing Care (UCC) (Active Comparator): UCC consists of a discharge recommendation to seek aftercare services at nearest treatment provider to where the patient lived. This service primarily consisted of outpatient group counseling.
  Interventions: Behavioral: UCC

INTERVENTIONS:
Behavioral: ACC — Weekly community based behavioral counseling and case management
  Arms: ACC + CM; Assertive Continuing Care (ACC)
Behavioral: CM — Weekly community based prize drawing opportunities contingent upon completed verifiable pro-social activities and clean urine and breath alcohol test results
  Arms: ACC + CM; Contingency Management (CM)
Behavioral: UCC — recommendation made by discharge counselor upon leaving residential treatment to attend nearest outpatient clinic.

SUMMARY:
Following discharge from residential treatment 324 adolescents are randomly assigned to Assertive Continuing Care with and without motivational incentives in a 2 x 2 factorial design. Clinical outcomes are assessed at 3, 6, 9, and 12 months post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Met DSM-IV diagnostic criteria for abuse or dependence on alcohol or another drug in the past year
* Been between the ages of 12 and 18 at the time of residential admission; and (c) resided in one of ten Illinois counties targeted for the intervention

Exclusion Criteria:

* left residential treatment prior to the seventh day
* did not return to a target county at discharge
* showed evidence of cognitive impairment that interfered with understanding of study instruments, procedures, or the informed consent process
* were deemed dangerous to themselves or others during treatment
* were a ward of child protective services and inaccessible for the intervention
* met DSM-IV criteria for pathological gambling
* were discharged to the state department of corrections
* were already participating in a treatment study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 342 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual)